CLINICAL TRIAL: NCT03573284
Title: Evaluating the Efficacy of Fractional Exhaled Nitric Oxide and Impulse Oscillometry in Patients With Cough Variant Asthma
Brief Title: Validity of Fractional Exhaled Nitric Oxide and Impulse Oscillometry in Patients With Cough Variant Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-HXNK-002
Record Dates: First submitted 2018-05-31; First posted 2018-06-29 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cough Variant Asthma
Keywords: cough variant asthma; chronic cough; fractional exhaled nitric oxide; impulse oscillometry; forced mid-expiratory flow
MeSH Terms: conditions — Cough-Variant Asthma; Chronic Cough | interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthma group (Experimental): Patients with chronic nonproductive cough for more than 8 weeks based on physician's opinion will be subjected to FeNO, impulse oscillometry(IOS) and pulmonary function. Receiver operating characteristic (ROC) curves to evaluate the clinical value of FeNO and small airways indices in CVA diagnosis. The optimal cutoff point for the level of FeNO and IOS is also determined.
  Interventions: Diagnostic Test: fractional exhaled nitric oxide(FeNO); Diagnostic Test: impulse oscillometry(IOS)

INTERVENTIONS:
Diagnostic Test: fractional exhaled nitric oxide(FeNO) — FeNO level was evaluated according to the American Thoracic Society (ATS)/ERS recommendations using a NIOX MINO analyzer (Aerocrine, Solna, Sweden) .Subjects were informed to deeply inhale NO-free air and immediately exhale in full via a mouthpiece at a constant flow rate (50 ml/s) for 10s.
Diagnostic Test: impulse oscillometry(IOS) — The patient take seats, body relax, make sure the mouthpiece is fully covered by mouth, then clip nose with both hands to cover both sides of the cheek, and then calm breathing 1 minutes, the computer is automatically collected data calculation and print out the measurement results.

SUMMARY:
The aim of the research is to evaluate the clinical value of fractional exhaled nitric oxide(FeNO) ,impulse oscillometry(IOS) and mid-expiratory flow (MEF) in patients with cough variant asthma.

DETAILED DESCRIPTION:
The present study has the following objectives:

to evaluate the relationship between BHR and mid-expiratory flow, to assess the diagnostic accuracy of fractional exhaled nitric oxide，impulse oscillometry and mid-expiratory flow in CVA with special regard to its discriminating value between CVA and other causes of a chronic cough, to estimate prognostic value of BHR and fractional exhaled nitric oxide (FeNO) count in predicting response to asthma treatment.

ELIGIBILITY:
Inclusion Criteria:

age 18-65 years old. Cough as the sole or predominant symptom lasting for at least 8 weeks, with no radiographic evidence of lung diseases.

Exclusion Criteria:

treatment of any oral corticosteroid in the last 4 weeks, and respiratory tract infection within 8 weeks.

smoking (min. 6 months) had asthma or other lung diseases, including obliterative bronchiolitis, bronchiectasis,and cystic fibrosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
the value of fractional exhaled nitric oxide(FeNO) in patients with cough variant asthma | at least 4 weeks of treatment
  FENO will be performed by using a hand-held portable machine (NIOX MINO, Aerocrine AB, Solna, Sweden) at a standard flow rate of 50 mL/s, in accordance with ATS/ERS recommendations.
the value of impulse oscillometry(IOS) in patients with cough variant asthma | at least 4 weeks of treatment
  R5-R20（respiratory resistance）is measure by Jaeger MasterScreen Pulmonary

SECONDARY OUTCOMES:
the value of forced mid-expiratory flow (MMEF) in patients with cough variant asthma | at least 4 weeks of treatment
  MMEF will be performed with a spirometer (Jaeger, Hoechberg, Germany) in accordance with the specifications and performance criteria recommended in the American Thoracic Society (ATS)/European Respiratory Society (ERS) Standardization of Spirometry
the value of BHR and fractional exhaled nitric oxide (FeNO) count in predicting response to asthma treatment | at least 4 weeks of treatment
  MCH bronchial provocation tests will be performed with the Jaeger APS Pro system.Provocative dose causing a 20% fall in FEV1(PD20) will be recorded, and BHR is defined as present if PD20≤0.48 mg. FENO is measure by a hand-held portable machine(NIOX MINO, Aerocrine AB, Solna, Sweden)
the relationship between BHR and mid-expiratory flow | at least 4 weeks of treatment
  BHR is measure by Jaeger APS Pro system.MMEF will be performed with a spirometer (Jaeger, Hoechberg, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hupeng, Principal Investigator — Southern Medical University, China
Locations (1):
- Huapeng Yu, Guangzhou, Guangdong, China